CLINICAL TRIAL: NCT03098355
Title: Anti-CD19/CD22 4th Generation CAR-T Cells (4SCAR19/22) Followed by Interleukin-2 Treating Pediatric Relapsed and Refractory B Cell Malignancies
Brief Title: Interleukin-2 Following 4SCAR19/22 T Cells Targeting Refractory and/or Recurrent B Cell Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The company did not offer the appropriate CART services.
Sponsor: Zhujiang Hospital (Other)
Collaborators: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: anti-CD19/22 CART Cells
Record Dates: First submitted 2017-03-26; First posted 2017-03-31 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2022-09

CONDITIONS: B-Cell Leukemia; B-Cell Lymphoma
Keywords: CART; CD19; CD22; Interleukin-2
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SCAR19/22 T cells and interleukin-2 (Experimental): Patients with resistant or refractory B cell acute lymphoblastic leukemia (ALL) or non-hodgkin's lymphoma (NHL) will receive CAR-T cells at a total dose of 0.5-5x10^6/kg and regular subcutaneous injection of interleukin-2 every other day for 2 weeks and then rest for 2 weeks for up to 6 months after their serum interleukin-6 levels returned to normal range from day 28 after CAR-T cell infusion.
  Interventions: Biological: 4SCAR19/22 T cells; Drug: Interleukin-2

INTERVENTIONS:
Biological: 4SCAR19/22 T cells — CD19/CD22-targeted 4th Generation CAR-T Cell (4SCAR19/22)
Drug: Interleukin-2 — Interleukin-2 of 250,000iu/m^2 every other day for 2 weeks and then rest for 2 weeks for up to 6 months.
  Other Names: IL-2

SUMMARY:
Clinical studies of CD19 CAR-T cells in the treatment of blood and lymphatic system tumors have achieved unprecedented successes. Because of the heterogeneity of the tumor, patients often carry CD19-negative tumor cell clones that express alternative target antigens (such as CD22, CD20 and CD123). In order to effectively eradicate all tumor clones and prevent recurrence, alternative tumor antigens besides CD19 are considered for CAR-T cell targeting. In this tudy, autologous T cells are genetically modified with 4th generation anti-CD19 and anti-CD22 CARs (4SCAR19/22) using lentiviral vectors. For safety consideration, the 4SCAR is engineered with an inducible caspase 9 self-withdrawal genetic design that allows for rapid elimination of the infused CAR-T cells. Interleukin-2 has been shown to boost immune response against leukemia cells. The serum interleukin-6 level will be monitored and when it returns to normal range by day 28 after CAR-T cell infusion, patients will receive subcutaneous injection of interleukin-2, and evaluated for 24 months for safety, efficacy and persistence of CAR T cells.

DETAILED DESCRIPTION:
Objectives:

1. Primary Outcome Measures:

   1. Evaluate the frequency and severity of adverse events, including, but not limited to, cytokine release syndrome (CRS) [ Time Frame: From date of dosing ( day 1 ) up to 50 weeks ]
   2. Evaluate grade 3 and higher toxicity rate of patients (toxicity possibly attributed to 4SCAR19/22 T cells)
   3. Evaluate the safety and effect of administration of 4SCAR19/22 T cells followed by interleukin-2 in treating pediatric patients with relapsed and refractory B cell malignancies.
2. Secondary:

   1. Evaluate Overall Complete Remission Rate (ORR).
   2. Evaluate overall response rate including complete remission (CR) and complete remission with incomplete blood count recovery (CRi) .
   3. Evaluate duration of remission (DOR).
   4. To evaluate the incidence and the treatment effect of cytokine release syndrome (CRS).
   5. To determine the expansion and functional persistence of 4SCAR19/22 T cells in the peripheral blood of patients and the correlation with antitumor effects;

Design:

1. In this single-center, open-label, nonrandomized, no control, prospective clinical trial, a total of 30 patients with resistant or refractory B cell acute lymphoblastic leukemia (ALL) or non-hodgkin's lymphoma (NHL) will be enrolled. Patients with ALL will be diagnosed according to bone marrow morphology, immunophenotype, cytogenetic and molecular examination. Patients with NHL will be diagnosed according to bone marrow morphology, biopsy pathology and imaging examination.
2. Peripheral blood mononuclear cells (PBMC) will be obtained by apheresis, and T cells will be activated and modified to express the 4SCAR-CD19/22 gene.
3. On Day -2 to -7, PBMC will be activated and enriched for T cells, which will be followed by 4SCAR-CD19/22 lentiviral transduction. The total culture time is approximately 5-7 days.
4. Patients will receive lymphodepleting chemotherapy composed of cyclophosphamide and fludarabine prior to cell infusion,
5. Participants will receive the CAR-T cells at a total dose of 0.5-5x10^6/kg.
6. Participants will receive regular subcutaneous injection of interleukin-2 of 250,000iu/m^2 every other day for 2 weeks and then rest for 2 weeks for up to 6 months after their serum interleukin-6 levels returned to normal range from day 28 after CAR-T cell infusion.
7. Patients will be monitored for toxicity including cytokine release syndrome, hematologic toxicities and B-cell aplasia, for response of their underlying malignancy and for CAR-T cell persistence in the blood, marrow and cerebral spinal fluid (CSF).

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory CD19+ B-cell lymphoma or leukemia.
2. Measurable disease.
3. Karnofsky/jansky score of 60% or greater.
4. ≥1 years old and ≤14 years.
5. Fertile females/males.
6. Expected survival>12 weeks.
7. Histologically confirmed as CD19/20-positive ALL/NHL and who meet one of the following conditions:

   1. Patients receive at least 2-4 prior combination chemotherapy regimens (not including single agent monoclonal antibody therapy) and fail to achieve CR.
   2. Recurrent disease and not eligible for allogeneic stem cell transplantation, and stable disease after therapy but refused further treatment.
   3. Disease recurrence after stem cell transplantation.
   4. Diagnosis as lymphoma, and refuse conventional treatment such as chemotherapy, radiation, stem cell transplantation and monoclonal antibody therapy.
8. Creatinine < 2.5 mg/dl.
9. Alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN.
10. Bilirubin < 2.0 mg/dl.
11. Adequate venous access for apheresis, and no other contraindications for leukapheresis.
12. Take contraceptive measures before recruit to this trial.
13. Written voluntary informed consent is given.

Exclusion Criteria:

1. A history of mental illness and poorly controlled.
2. Patients with symptoms of central nervous system.
3. Suffering severe cardiovascular or respiratory disease.
4. Accompanied by other malignant tumor.
5. Known human immunodeficiency virus (HIV) infection.
6. Active and/or severe infection (e.g. tuberculosis, sepsis and opportunistic infections, active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection).
7. Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the patient.
8. Taking immunosuppressive agents within 1 week due to organ transplantation or other disease which need long-lasting administration.
9. Patients that do not consent to tissue and blood sample collection and storage in a biobank.
10. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed 48 hours before infusion.
11. Pregnancy and nursing females.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the frequency and severity of adverse events including, but not limited to, cytokine release syndrome (CRS) | From date of dosing ( day 1 ) up to 50 weeks
  b)Evaluate grade 3 and higher toxicity rate of patients (toxicity possibly attributed to 4SCAR19/22 T cells)

CONTACTS AND LOCATIONS:
Overall Officials: Li-hua Yang, Ph.D., Principal Investigator — Southern Medical University, China; Lung-Ji Chang, Ph.D., Study Director — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No